CLINICAL TRIAL: NCT03395613
Title: Prophylactic Use of a Negative Pressure Incision Management System in Infrainguinal Vascular Surgery - A Multicentre Randomized Controlled Trial
Brief Title: Negative Pressure Incision Management System in Infrainguinal Vascular Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Alireza Daryapeyma, MD PhD, Principal Investigator, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ADaryapeyma
Record Dates: First submitted 2017-12-27; First posted 2018-01-10 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Surgical Site Infection

STUDY DESIGN:
Intervention Model Description: Preoperative randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard management (No Intervention): Standard sterile gauze dressing on surgical groin wound.
- NPWT management (Experimental): Negative Pressure Wound Therapy dressing on surgical groin wound.
  Interventions: Device: NPWT

INTERVENTIONS:
Device: NPWT — Negative pressure wound thearpy on closed surgical wounds
  Other Names: Prevena
  Arms: NPWT management

SUMMARY:
Negative pressure wound therapy (NPWT) has been used in treating postoperative SSI with encouraging results and is now an accepted element in the arsenal of tools for treating these complications. The concept of applying NPWT to closed surgical wounds as a preventive measure is relatively new but draws on the inherent properties of the method which could theoretically lead to reduced seroma formation, wound dehiscence, increased capillary circulation and consequently better wound healing and fewer SSI.

Given the incidence and the consequences of SSI in infrainguinal vascular procedures any appreciable decrease in the burden of these complications could have profound benefits for patients and healthcare facilities. As to date, there are no published data from randomized controlled trials investigating the effectiveness of this prophylactic measure.

The aim of this study is to assess the effect of NPWT applied to closed surgical wounds directly after skin closure compared to standard sterile gauze dressing in reducing the incidence and severity of postoperative SSI in infrainguinal surgical wounds in patients undergoing elective, open vascular surgery.

DETAILED DESCRIPTION:
Intervention and Surveillance:

The groin incisions in the intervention group will have NPWT dressing, applied under sterile conditions in the operating room. The NPWT will remain on the patient until postoperative day 7 or earlier if the vacuum seal is broken for any reason. If the NPWT is removed earlier than 7 days, a sterile gauze dressing will be applied to the incision.

The control group will receive a sterile gauze dressing, applied under sterile conditions in the operating room. The dressing van if needed be changed under sterile conditions at the ward on the second postoperative day. The dressing will remain on the patients until postoperative day 7. The dressing may be changed (by a research nurse or the attending surgeon), under sterile conditions if needed during the 8-day period.

After the initial 8-day period, patients in both groups will be supplied with sterile gauze dressings for an additional 6 days during which dressing changes may be carried out under sterile conditions.

All groin incisions will be examined, evaluated and categorized by a qualified research nurse or the attending surgeon, who will be blinded to the initial treatment modality, on the seventh postoperative day, 30 days postoperative and again after three months. Wound cultures will be taken (when possible) if the ASEPSIS score at any one of the three examinations is equal to, or exceeds 21 points.

Preoperative preparations will be the same for both groups. All patients will receive three doses (one pre- and two postoperative) of antibiotic prophylaxis on the day of the operation. Groin incisions will be closed with subcutaneous and intracutaneous monofilament absorbable sutures.

All patients will be asked to respond to the 36-Item Short Form Health Survey (SF-36) and the European Quality of life - Five dimensions (EQ-5D) questionnaires at the time of inclusion and at the one month follow up visit. The Wound QoL (Swedish) questionnaire will be presented to the patients at the one-week follow up.

Primary Endpoint:

• Postoperative SSI within 30 day, classified according to the scoring method ASEPSIS (Additional treatment,Serous discharge, Erythema, Purulent exudates, Separation of the deep tissues, Isolation of bacteria and in-patient Stay) and graded using the Samson classification (Grade I-V), confirmed by positive identification of the infectious agent.

Secondary Endpoints:

Postoperative SSI within 90 days, classified according to the scoring method ASEPSIS (Additional treatment,Serous discharge, Erythema, Purulent exudates, Separation of the deep tissues, Isolation of bacteria and in-patient Stay) and graded using the Samson classification (Grade I-V), confirmed by positive identification of the infectious agent.

* Antibiotic prescriptions for skin and soft tissue infections within 90 days postoperatively.
* Postoperative SSI within 90 days requiring surgical revision.
* Adverse events directly related the NPWT dressing leading discontinuation of treatment.
* Major lower limb amputation and/or mortality within 90 days postoperatively.
* Changes in reported functionality and quality of life during the 30 day postoperative period.
* Assessment of healthcare related costs within 30 days postoperatively.

Based on previous studies the incidence of postoperative groin SSI is 30-35%. Recent studies using NPWT have shown a reduction in incidence of 50% or more.

Using a sample size calculator (Sealed Envelope Ltd., Clerkenwell Workshops, London EC1R 0AT, UK) for binary outcome superiority trials with an alpha level of 0.05 for 80% power and an estimated incidence reduction from 30% to 10% using NPWT a sample size of 59 patients in each arm and a total sample size of 118 is required.

Randomization will occur once the skin incision has been closed. In cases of bilateral groin incision the right groin will be randomized and the left allocated the other arm of the trial. The surgeons, the operating room personnel and the investigators evaluating the outcome will not be blinded to the intervention.

Missing data will be treated based on the type data missing. In cases where missing data will affect the primary outcome the cases wil be deleted but accounted for in the final report.

Statistical Analysis Plan:

The data from each patient will be analysed using appropriate statistical methods for categorical and continuous and comparative analysis in respect to risk factors and outcome, both primary and secondary as previously defined. Absolute risk increase or reduction, as well as numbers needed to treat for NPWT use will be reported.

Analysis of primary outcomes will be done based on the intention to treat principle. Student's t-test and Pearson's chi-square or Fisher's exact test for continuous and categorical data, respectively. In cases where bilateral incisions are planned, the right groin will be randomized and the left will receive the alternate treatment. For subjects lost to follow up, the last recorded follow up/outcome will be recorded as their final outcome.

Analysis of secondary outcome data will be done according to normal distribution of data whrereby non-normally distributed data will be analysed using the Mann-Whitney U-test.

All tests will be 2-sided and P ≤ 0.05 will be considered statistically signinficant for all tests.

The statistical analyses will be done using SPSS version 23 (IBM, Armonk, NY, USA).

All patients will be asked to respond to the 36-Item Short Form Health Survey (SF-36) and European Quality of life - Five dimensions (EQ-5D) and Wound QoL questionnaires at the time of inclusion and at the one month follow up visit.

The data from these questionnaires will be stratified and analysed using appropriate statistical methods.

Ethical considerations:

General regulations The study will be performed in accordance with the declaration of Helsinki as revised at the 64th WMA General Assembly in Fortaleza, Brazil, October 2013. Approval of the study protocol has been obtained from the Regional Ethics Committee.

Informed consent Prior to enrolment all patients will receive written and oral information about the study. The patients will only be included after obtaining written and informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years.
2. The clinical criterion for study entry is elective:

   a. Open infrainguinal vascular surgery for peripheral arterial disease

   i. Thrombendarterectomy (TEA) ii. Bypass surgery with vein or synthetic graft
3. Patients on whom complete seal of NPWT can be maintained during the first 24 hours after operation.

   -

Exclusion Criteria:

1. All emergency cases.
2. Infrainguinal endovascular procedures.
3. Pre-existing groin infections.
4. Sensitivity/allergy to materials used in NPWT dressing.
5. Patients on whom an adequate and complete seal of NPWT dressing cannot be obtained.
6. Unwillingness to participate. -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative surgical site infection (SSI) within 30 days. | 30 days
  SSI classified according to the scoring method ASEPSIS (Additional treatment,Serous discharge, Erythema, Purulent exudates, Separation of the deep tissues, Isolation of bacteria and inpatient Stay) and graded using the Samson classification (Grade I-V), confirmed by positive identification of the infectious agent.

SECONDARY OUTCOMES:
Postoperative SSI within 90 days | 90 days
  SSI classified according to the scoring method ASEPSIS (Additional treatment,Serous discharge, Erythmea, Purulent exudates, Separation of the deep tissues, Isolation of bacteria and inpatient Stay) and graded using the Samson classification (Grade I-V), confirmed by positive identification of the infectious agent.
Antibiotic prescriptions for skin and soft tissue infections within 90 days postoperatively. | 90 days
Postoperative SSI within 90 days requiring surgical revision. | 90 days
Adverse events directly related the NPWT dressing leading discontinuation of treatment. | 7 dats
  Death due to procedural complications
  * Vascular complications
  * Severe or life-threatening bleeding
  * Limb loss
  * TIA/stroke or myocardial infarction
  * Allergic skin reactions
  * Device related skin damage e.g. abrasions, blisters or wounds
Major lower limb amputation and/or mortality within 90 days postoperatively. | 90 days
Changes in reported quality of life during the 30 day postoperative period. | 30 days
  Changes in QoL assessment questionnaires (SF-36 and EQ-5D) preoperatively and 30 days postoperative.
Assessment of healthcare related costs within 30 days postoperatively. | 30 days
Assessment of quality of life during the first seven day period after operation | 7 days
  The Wound QoL questionnaire will help assess QoL during the period that the NPWT device (Prevena) will be used in patients randomized to the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Daryapeyma, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska university Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vriesendorp TM, Morelis QJ, Devries JH, Legemate DA, Hoekstra JB. Early post-operative glucose levels are an independent risk factor for infection after peripheral vascular surgery. A retrospective study. Eur J Vasc Endovasc Surg. 2004 Nov;28(5):520-5. doi: 10.1016/j.ejvs.2004.08.006. PMID 15465374
- [Background] Cater JE, van der Linden J. Simulation of carbon dioxide insufflation via a diffuser in an open surgical wound model. Med Eng Phys. 2015 Jan;37(1):121-5. doi: 10.1016/j.medengphy.2014.07.011. Epub 2014 Aug 5. PMID 25103346
- [Background] Turtiainen J, Saimanen EI, Makinen KT, Nykanen AI, Venermo MA, Uurto IT, Hakala T. Effect of triclosan-coated sutures on the incidence of surgical wound infection after lower limb revascularization surgery: a randomized controlled trial. World J Surg. 2012 Oct;36(10):2528-34. doi: 10.1007/s00268-012-1655-4. PMID 22618956
- [Result] Vogel TR, Dombrovskiy VY, Carson JL, Haser PB, Lowry SF, Graham AM. Infectious complications after elective vascular surgical procedures. J Vasc Surg. 2010 Jan;51(1):122-9; discussion 129-30. doi: 10.1016/j.jvs.2009.08.006. Epub 2009 Dec 2. PMID 19954920
- [Result] Kent KC, Bartek S, Kuntz KM, Anninos E, Skillman JJ. Prospective study of wound complications in continuous infrainguinal incisions after lower limb arterial reconstruction: incidence, risk factors, and cost. Surgery. 1996 Apr;119(4):378-83. doi: 10.1016/s0039-6060(96)80135-8. PMID 8644000
- [Result] de Lissovoy G, Fraeman K, Hutchins V, Murphy D, Song D, Vaughn BB. Surgical site infection: incidence and impact on hospital utilization and treatment costs. Am J Infect Control. 2009 Jun;37(5):387-397. doi: 10.1016/j.ajic.2008.12.010. Epub 2009 Apr 23. PMID 19398246
- [Result] Kuy S, Dua A, Desai S, Dua A, Patel B, Tondravi N, Seabrook GR, Brown KR, Lewis BD, Lee CJ, Kuy S, Subbarayan R, Rossi PJ. Surgical site infections after lower extremity revascularization procedures involving groin incisions. Ann Vasc Surg. 2014 Jan;28(1):53-8. doi: 10.1016/j.avsg.2013.08.002. Epub 2013 Nov 1. PMID 24189008
- [Result] Krizek TJ, Robson MC. Evolution of quantitative bacteriology in wound management. Am J Surg. 1975 Nov;130(5):579-84. doi: 10.1016/0002-9610(75)90516-4. No abstract available. PMID 1106243
- [Result] Arbeit RD, Dunn RM. Expression of capsular polysaccharide during experimental focal infection with Staphylococcus aureus. J Infect Dis. 1987 Dec;156(6):947-52. doi: 10.1093/infdis/156.6.947. PMID 3680994
- [Result] Garibaldi RA, Cushing D, Lerer T. Risk factors for postoperative infection. Am J Med. 1991 Sep 16;91(3B):158S-163S. doi: 10.1016/0002-9343(91)90362-2. PMID 1928157
- [Result] Chang JK, Calligaro KD, Ryan S, Runyan D, Dougherty MJ, Stern JJ. Risk factors associated with infection of lower extremity revascularization: analysis of 365 procedures performed at a teaching hospital. Ann Vasc Surg. 2003 Jan;17(1):91-6. doi: 10.1007/s10016-001-0337-8. Epub 2003 Jan 15. PMID 12522701
- [Result] Anderson DJ. Surgical site infections. Infect Dis Clin North Am. 2011 Mar;25(1):135-53. doi: 10.1016/j.idc.2010.11.004. PMID 21315998
- [Result] Lee ES, Santilli SM, Olson MM, Kuskowski MA, Lee JT. Wound infection after infrainguinal bypass operations: multivariate analysis of putative risk factors. Surg Infect (Larchmt). 2000 Winter;1(4):257-63. doi: 10.1089/109629600750067183. PMID 12594881
- [Result] Dosluoglu HH, Loghmanee C, Lall P, Cherr GS, Harris LM, Dryjski ML. Management of early (<30 day) vascular groin infections using vacuum-assisted closure alone without muscle flap coverage in a consecutive patient series. J Vasc Surg. 2010 May;51(5):1160-6. doi: 10.1016/j.jvs.2009.11.053. Epub 2010 Mar 31. PMID 20356703
- [Result] Weed T, Ratliff C, Drake DB. Quantifying bacterial bioburden during negative pressure wound therapy: does the wound VAC enhance bacterial clearance? Ann Plast Surg. 2004 Mar;52(3):276-9; discussion 279-80. doi: 10.1097/01.sap.0000111861.75927.4d. PMID 15156981
- [Result] Matatov T, Reddy KN, Doucet LD, Zhao CX, Zhang WW. Experience with a new negative pressure incision management system in prevention of groin wound infection in vascular surgery patients. J Vasc Surg. 2013 Mar;57(3):791-5. doi: 10.1016/j.jvs.2012.09.037. Epub 2013 Jan 9. PMID 23312938
- [Result] Hyldig N, Birke-Sorensen H, Kruse M, Vinter C, Joergensen JS, Sorensen JA, Mogensen O, Lamont RF, Bille C. Meta-analysis of negative-pressure wound therapy for closed surgical incisions. Br J Surg. 2016 Apr;103(5):477-86. doi: 10.1002/bjs.10084. PMID 26994715
- [Result] Daryapeyma A, Hammar U, Wahlgren CM. Incidence of Healthcare Associated Infections After Lower Extremity Revascularization Using Antibiotic Treatment as a Marker. Eur J Vasc Endovasc Surg. 2016 May;51(5):690-5. doi: 10.1016/j.ejvs.2015.12.016. Epub 2016 Feb 20. PMID 26905472
- [Derived] Daryapeyma A, Nilsson O, Pettersson J, Stackelberg O, Torbjornsson E, Hultgren R. Prophylactic use of incisional negative pressure wound therapy for groin incisions in vascular surgery: randomized clinical trial. BJS Open. 2025 May 7;9(3):zraf059. doi: 10.1093/bjsopen/zraf059. PMID 40500745